CLINICAL TRIAL: NCT02515851
Title: A Randomized, Double-blind Controlled Trial of Bupivacaine Extended-release Liposome Injection for Postsurgical Analgesia in Patients Undergoing Open-reduction Internal Fixation of the Distal Radius
Brief Title: Postsurgical Bupivacaine Extended-release Liposome Injection for Open-reduction Internal Distal Radius Fixation.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to find sufficient drug naive patients
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, David Seligson, Principal investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-086
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Group (Active Comparator): Group that receives actual liposomal bupivacaine injections
  Interventions: Drug: Exparel
- Placebo Group (Placebo Comparator): Group that receives placebo injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exparel
  Other Names: Liposomal Bupivacaine
  Arms: Active Group
Drug: Placebo
  Arms: Placebo Group

SUMMARY:
For patients undergoing open-reduction internal-fixaton (ORIF) of isolated distal radius fractures, administration of 66.5 mg of liposomal bupivacaine to operative field may decrease the need for post-operative narcotic pain medication.

DETAILED DESCRIPTION:
TITLE OF THE RESEARCH PROJECT A randomized, double-blind controlled trial of bupivacaine extended-release liposome injection for post-surgical analgesia in patients undergoing open-reduction internal fixation of the distal radius.

PROJECT SUMMARY For patients undergoing open-reduction internal-fixaton (ORIF) of isolated distal radius fractures, administration of 66.5 mg of liposomal bupivacaine to operative field may decrease the need for post-operative narcotic pain medication.

STATEMENT OF THE PROBLEM Patients undergoing open-reduction internal-fixation (ORIF) of isolated distal radius fractures experience significant post-operative pain, most commonly mitigated by the use of narcotic painkillers. Among other issues, prolonged use of narcotic painkillers can lead to dependence and abuse. This potentially leads to post-operative narcotic seeking habits of adult orthopedic trauma patients.

THEORETICAL FRAMEWORK There is much research supporting that administration of liposomal bupivacaine is an effective post-surgical analgesic. The investigators' hypothesis is that 66.5 mg of liposomal bupivacaine injected at the operative field will decrease the need for post-operative narcotics, and will therefore reduce the risk of dependence and abuse.

RESEARCH OBJECTIVE

-Assess the potential benefit of single-dose liposomal bupivacaine (Exparel) in the treatment of post-operative pain following open-reduction internal-fixation of isolated distal radius fractures.

METHODOLOGY Patients admitted to University of Louisville Hospital with isolated distal radius fractures requiring ORIF will be eligible. Exclusion criteria will be as follows: 1) patients who have received narcotic pain medication within the past 6 months as confirmed by Kasper reporting 2) Patients compartment syndrome or acute carpal tunnel syndrome requiring surgical decompression 3) Patients with prior history of ipsilateral wrist surgery.

Randomization will be performed using sealed envelopes, and each patient will be assigned a number that corresponds to either an Exparel 266mg solution (20 ml Exparel 1.3% plus 40ml of injectable saline) verses a 60ml placebo control injection (20ml inert liposomal suspension used in the manufacturing of Exparel without bupivacaine plus 40ml injectable saline) to be provided by Pacira. If inert liposomal solution is not a viable option, blinded/opaque syringes (either provided by Pacira (preferable ) or created by unblinded personnel) will be used to dispense 60 mL of sterile saline. The corresponding solution will be known to the participating, unblinded pharmacists who will provide the solutions and keep participant records, and not to the surgeons.

The amount of narcotic pain medication used in the recovery room and during the hospital admission will be recorded. Patients will also be provided study logs to record their daily usage of prescribed pain medication once discharge home. Follow-up phone calls will be made to each patient 72 hours post-operatively, and the amount of narcotic tablets used will be recorded. Patients will then be seen in the clinic 1 week postoperatively, and the total narcotic pain medication usage will again be documented. Passive wrist range of motion (ROM) tolerance and overall satisfaction will also be assessed at this visit. Demographic data including age, gender and handedness will be recorded for each patient. The primary outcome measure will be the total post-operative narcotic pain medication use. Secondary outcome measures will be passive wrist ROM, and overall satisfaction.

All subjects will be treated ethically. This includes true informed consent, explanation of the study by a co-investigator, and time to ask questions about the study. Patient intake data will be kept on paper forms initially and kept in a desk behind a locked research office in the department of orthopaedics that is accessible only to staff. This data will be entered into a password protected computer in the same office and the papers will then be shredded. Once feasible, all PHI will be removed from the data set. A key for the PHI will be in a separate excel file on this same computer.

PLAN FOR ANALYSIS OF RESULTS To detect a 30% difference in narcotic pain medication requirement, a Cohen's d = 0.4 (small/medium effect) will be required.

TIMETABLE The study will begin once IRB approval is obtained and will continue for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Isolated distal radius fracture

Exclusion Criteria:

* No Access to a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Seligson, MD, Principal Investigator — University of Louisville

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Group: Group that receives actual liposomal bupivacaine injections
  Exparel
- Placebo Group: Group that receives placebo injections
  Placebo
Period: Overall Study
Arm/Group | Active Group | Placebo Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group | Placebo Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Pain Medication Usage
Description: the amount of pain medication used in the three days following surgery.
Time Frame: three days
Population: Data were not collected
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Total Narcotic Pain Medication Usage
Description: The total narcotic pain medication usage for 1 week after surgery
Time Frame: 7 days after surgery
Population: Data were not collected
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Passive Wrist Range of Motion
Description: Wrist range of motion possible when surgeon moves the wrist between 0 and 180 degrees.
Time Frame: 7 days after surgery
Population: Data were not collected
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Over Satisfaction
Description: Patients will rate satisfaction with their surgery and recovery on a 1 to 10 scale with 1 being the lest and 10 being the most satisfied.
Time Frame: 7 days after surgery
Population: Data were not collected
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Active Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes